CLINICAL TRIAL: NCT00647257
Title: The Effect of Losartan on Atrial Fibrillation and Pacemaker Dependence in Sick Sinus Syndrome (SSS) Patients Receiving Physiological Pacemaker - A Prospective, Randomized, Multicenter Study in Taiwan
Brief Title: The Effect of Losartan on Atrial Fibrillation (AF) Burden and Pacemaker Dependence in Patients With Sick Sinus Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Kwo-Chang Ueng, Chung Shan Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COZ-002-00-28SEP2007
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2010-04-01 (Estimated); Status verified 2010-03

CONDITIONS: Atrial Fibrillation
Keywords: Sick Sinus Syndrome; Atrial Fibrillation; Pacemaker
MeSH Terms: conditions — Atrial Fibrillation; Sick Sinus Syndrome | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Losartan
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Losartan — Patients, aged 20 to 80 years, with SSS will be enrolled and randomly assigned to the Losartan 100mg add on physiological atrial-based pacing or physiological atrial-based pacing alone treatment arm.
  Arms: A
Drug: Placebo — Patients, aged 20 to 80 years, with SSS will be enrolled and randomly assigned to the Placebo add on physiological atrial-based pacing or physiological atrial-based pacing alone treatment arm.
  Arms: B

SUMMARY:
This is a an investigator-initial, multicenter, open-label, randomized, parallel-group comparative study to evaluate the effect on the incidence of AF and pacemaker dependence in SSS patients receiving physiological atrial-based pacing alone or adding losartan 100mg to physiological atrial-based pacing treatment. The duration of the study will be approximately 13 months, comprising 4-week pre-study period, and 12-month treatment period.

DETAILED DESCRIPTION:
Sick sinus syndrome is a common indication for permanent cardiac pacing in the community. It results from disordered impulse generation within the sinus node or impaired conduction of the impulse to the surrounding atrial tissue, thus leading to the clinical manifestation of bradycardia. In patients with SSS, AF frequently develops after pacemaker implantation,and progresses to persistent AF over long term follow up.

The occurrence of AF have been shown to be an independent predictor for major cardiovascular events in SSS patients receiving physiologic pacing. Recent prospective clinical trials have demonstrated that physiologic pacing mode reduces the risk of AF compared to single chamber ventricular pacing in patients with SSS. However, the effectiveness of physiologic pacing in reducing the incidence of AF in patients with sinus node dysfunction is still incomplete.

One recent clinical study had reported that 68% of SSS patients with a DDDR pacemaker have atrial tachyarrhythmias detected by the pacemaker devices at median 718 days follow-up. Modern pacemakers have diagnostic features that permit the detection and storage of information about the date, time of onset, and duration of multiple, sequential episodes of atrial tachyarrhythmias. Since a high percentage of AF episodes may be asymptomatic, AF "burden" have been used as surrogate end points. Prolonged P wave, shortened refractoriness, or remarkably abnormal conduction disturbances in the presence of prolonged refractoriness limit the effectiveness of standard physiologic pacing in AF prevention. This could explain, at least in part, the tendency of SSS to develop AF as a part of its natural history. Clinical electrophysiology has focused the attention on the electrophysiological and structural properties of the atrial muscle in patients with SSS: shortened and inhomogeneous refractoriness and local and regional conduction slowing, as well as prolonged intra- and inter-atrial conduction disturbances, are well described as increased interstitial fibrosis associated with the genesis of AF.

A growing body of evidences has shown that inhibition of the renin-angiotensin system can prevent the promotion of AF by suppressing the development of atrial fibrosis and structural remodeling. At present, the influence of a treatment target aiming on altered fibrosis and structural substrate in patients with SSS is not yet known. One striking result of the losartan intervention for endpoint reduction in hypertension (LIFE) study was that new-onset AF and associated stroke were significantly reduced by losartan- compared to atenolol-based antihypertensive treatment with similar blood pressure reduction.

The relative risk of new-onset AF in losartan group is 0.67 compared to atenolol group (i.e.; 33% risk reduction) Therefore, there is every reason to believe that blocking the renin-angiotensin pathway with angiotensin II type 1 receptor blockade would have positive influence on AF burden in this clinical setting. Recently, enalapril has been reported to prevent rapid atrial pacing (4 weeks)-induced interstitial fibrosis and fatty degeneration of the sinus node and to improve sinus node function in canine model, supporting the important role of structural changes of sinus node in the regulation of sinus node function. This possibility supporting therapeutic interventions using RAS inhibitors forms an attractive theoretical basis for interventions to reverse SND in such patients.

In support of these hypotheses, the present study was undertaken to determine whether selective angiotensin II type 1 receptor blockade with high dose losartan was effective in reducing AF burden, pacemaker dependence, shortening of sinus node recovery time, hsCRP, and NT-pro BNP, and associated cardiovascular events in SSS patients receiving physiologic pacing.

In this study, all pacemakers are standard rate-adaptive dual chamber pacemakers:

Medtronic Kappa 900 or Versa. At implantation, all patients were programmed to DDI mode at 50 ppm to minimize the ventricular pacing. All patients had the atrial tachyarrhythmia detection feature programmed "on" after pacemaker implantation. This feature provides information on the date, time of onset, and duration of the first 15 consecutive episodes of an atrial tachyarrhythmia. This information can be retrieved during follow-up visits using the pacemaker programmer.Patients were evaluated every 3 months after pacemaker implantation. At each visit, the atrial tachyarrhythmia diagnostic data were retrieved. Each episode classified as an atrial tachyarrhythmia was reviewed by one of the investigators. False-positive detections of AF due to oversensing were excluded using specific rules developed in the course of previous clinical trials. On review of the beat-to-beat intervals stored in the diagnostic counters during an episode classified as AF, far-field oversensing was defined if

1. Long intervals between successive detected atrial events were paced and short intervals were sensed; or
2. The difference between the first, third, fifth, and seventh atrial intervals and the second, fourth, sixth, and eighth intervals was > 150 beats/min; or
3. The sum of the long and short interatrial intervals was equal to the interatrial intervals recorded before or after termination of the episode.

The atrial tachycardia detection feature in the Medtronic Kappa 900 or Versa was used for AF detection in this study. This feature has been reported to have a high sensitivity and specificity for the detection of atrial tachyarrhythmias. All atrial leads were bipolar. The atrial sensitivity was programmed to 0.5 mV, which is the standard clinic protocol. The programming parameters for AF detection included a post-ventricular atrial blanking period of 150 msec, a tachycardia detection rate of 180 beats/min, the number of beats for atrial tachycardia detection of 200, the number of beats for tachycardia termination of 10, and the diagnostic arrhythmia counter was frozen in order to collect information on the first 15 tachycardia episodes. These parameters were selected to optimize the detection of AF and to reduce the likelihood that nonsustained AF would fill the diagnostic counters. AF episodes < 1 minute in duration were not detected as an episode of AF. To maximize collection of sequential episodes of AF, the atrial electrogram storage feature was not used. In the Kappa 900 or Versa, an electrogram can be retrieved for the first episode of AF detected (if the episode occurs within a programmable time) and, in these cases, the electrogram was reviewed to ensure appropriate classification of AF.

Sustained AF was defined as an atrial tachyarrhythmia with an atrial rate > 250 beats/min and duration > 1 minute. The atrial rate was determined based on review of the interatrial intervals stored in the device diagnostics during each episode.

AF burden was defined as the quantity of AF documented during the follow-up period and expressed as a portion of the follow-up period (hours/day). When the event counters were filled, AF burden was calculated as the total duration of AF during the time required to fill the counters.

Permanent AF was defined as AF present at two consecutive visits and an AF burden of 24 hours/day between those visits.

CSNRT at pacemaker implant and each visit :

The corrected sinus node recovery time (CSNRT) was assessed at CLs of 600, 500 and 400 ms after a 30-second pacing train from the atrial lead. The measurement of CSNRT was repeated 3 times, and averaged. Atrial-based pacemaker dependence Pacemaker dependency was defined as the absence of escape or intrinsic rhythm for at least 30 seconds after gradual slowing of the pacing rate to 30 beats/min. Pacemaker dependency was examined every 3 months. Measurement of Intrinsic Heart Rate Pacing system follow-ups, including measurements of pacing/sensing characteristics, lead impedance, and surveillance of battery status were performed every 3 months in each patient. Endocardial atrial and ventricular electrograms were recorded via a programmer with the pacing mode temporarily set to AAI at a lower rate of 30 beats/min. A temporary programmable function that allows markers to appear on the programmer's electrocardiographic recording, corresponding to spontaneous events sensed by the pulse generator, was used to measure the rate of intrinsic or escape rhythms.

Pacing rate was manually step-downed to 30 beats/min in every 10 beats/min from the lower pacing rate, and intrinsic or escape rhythms were checked at each pacing rate. A fixed pacing rate of 30 beats/min following the gradual decrease was maintained for at least 30 seconds to allow the emergence of intrinsic or escape rhythms.

Approximately 220 male and female patients, aged 20 to 80 years, with SSS will be enrolled and randomly assigned to the losartan add on physiological atrial-based pacing or physiological atrial-based pacing alone treatment arm. The sample size was calculated to provide the study with 80% power for a two-sided alpha level of 0.05. Assuming a 33% reduction of AF incidence rate in the losartan group compared with physiological pacing only group after 1 year after randomization. Based on these assumptions, the total sample size required was estimated to be 100 patients in each arm. Thus we need to enroll 220 eligible cases.

Study medication (losartan) will be in tablet form. Patients randomized to the losartan arm will receive 50 mg once a day for 2 weeks, patients will then be up-titrated to 50 mg of losartan twice a day following the first 2-week therapy. Each patient will be assessed following 4 weeks of losartan therapy at this dose. If the patient is well tolerated for this dose they will be maintained on it for the remaining time of the study. If they are unable to tolerate this target dose they will be permitted to down-titrate and continue on the highest tolerated dose. Only those patients able to tolerate at least the lowest dose of losartan will be permitted to continue on study until the end of study period.

Normotensive patients who weigh less than 50 kg, or who are aged over 70 years will receive 25 mg/day for the first 2 weeks, then increase to 50 mg/day, with the aim of reaching 100 mg/day for the rest of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing to sign informed consent form.
* Men or women ≧ 20 and ≦ 80 years of age.
* Symptomatic bradycardia < 40 beats/min or symptomatic QRS pauses of more than two seconds.
* Normal AV conduction (PQ interval ≦ 220 ms for patients≦ 70 years and a PQ interval ≦ 260 ms for patients >70 years), and no bundle branch block (QRS width < 120 ms)

Exclusion Criteria:

* Patient has history of known intolerance, contraindication or hypersensitivity to losartan.
* 1st, 2nd or 3rd AV block
* Permanent or therapy refractory AF
* Blood pressure > 250/120 mmHg at visit 1.
* Heart Failure acc. NYHA III or IV
* Myocardial infarction less than 6 months before pacemaker implant (visit 1)
* Cerebral disease or stroke less than 6 months before pacemaker implant (visit 1)
* Hypertrophic obstructive cardiomyopathy
* Symptomatic hypo- or hyperthyroidism
* Cardiogenic shock
* Women who are pregnant or lactating.
* Unstable angina pectoris
* Patients under 20 years of age
* Patients involved in other studies
* Systolic pressure < 100 mmHg at the visit 1
* Reduced expectancy of life due to other diseases
* Patients who cannot attend follow-up visits regularly
* Patient has clinically important abnormal laboratory findings at the visit 1 local laboratory screen including: Serum creatinine > 2.5 mg/dL; Serum potassium < 3.5 or > 5.7 eEq/L; SGOT/SGPT (ALT/AST) > 3 times of the upper normal limits; Blood hemoglobin (males & females < 10 g/dL)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients who developed AF burden by pacemaker telemetry and developed permanent AF | 12-month study period(2-week + 2-week + 4-week + 4-week + 3-month + 3-month + 3-month)

SECONDARY OUTCOMES:
The time to first occurrence of AF lasting for at least 1 minute after pacemaker insertion, and the AF burden over time measured as the portion of AF per day (in hours/day) | 12-month study period(2-week + 2-week + 4-week + 4-week + 3-month + 3-month + 3-month)

CONTACTS AND LOCATIONS:
Overall Officials: Kwo-Chang Ueng, MD; PhD, Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan